CLINICAL TRIAL: NCT02931656
Title: Acute Effects of an Aquatic Physical Exercise on Glycemic Control of Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Collaborators: Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, José Roberto da Silva Junior, Professor Fernando Figueira Integral Medicine Institute, Professor Fernando Figueira Integral Medicine Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1111-1188-1100
Record Dates: First submitted 2016-09-28; First posted 2016-10-13 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Diabetes, Gestational
Keywords: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Aquatic Therapy; Hydrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GDM aquatic exercise (Experimental): GDM Diagnosis criteria accordance with to IADPSG / WHO
  Interventions: Other: Aquatic exercise
- Control Group aquatic exercise (Active Comparator): No change in blood glucose levels Group, investigated between 24-28 weeks of gestation.
  Interventions: Other: Aquatic exercise

INTERVENTIONS:
Other: Aquatic exercise — The aquatic exercise program will be under the professional guidance of a physiotherapist, with water at a temperature of around 26 to 28°C. The exercise sessions will be executed following the steps: 1) Heating (stretching and flexibility, static method, during 5'); 2) Aerobic exercise (running, displacements and combined movements of arms and legs, with 1minute interval, to 1minute activity and of during 20') 3) Spot exercises (strength / endurance of the upper and lower limbs and abdomen, using the resistance of water for 15') 4) Relaxation (slow walks for 5'). During the sessions of exercises the pregnant women will have heart rate monitored by the frequency meter (Polar Electro OY) to control the intensity of the exercises that will focus on the range of moderate intensity.
  Other Names: Water aerobics; Hydrotherapy

SUMMARY:
Gestational diabetes mellitus (GDM) is increasing worldwide and has been associated with adverse perinatal outcomes and high risk for chronic disease both for the mother and for the child. Physical exercise is feasible to diabetic pregnant women and contributes to a better glycemic control and to decrease adverse perinatal outcomes. However there are no studies assessing the effects of aquatic physical exercise on GDM control.

DETAILED DESCRIPTION:
The study will be conducted at Institute of Medicine Professor Fernando Figueira (IMIP), Brazil. The patients will be included in the study by consent after an explanation of the study goals. Women will be considered eligible for enrollment if they fulfill all the inclusion criteria and none of the exclusion criteria. Sample size was calculated with the aim of reducing glucose levels by 20% in intervention GDM group. A power of 80% and a level of significance of 5% was accepted and the calculated sample size in each arm was 30 patients. Assuming a drop out of 20%, 72 pregnant women will be included in the study. 36 gestational diabetics and and 36 normoglycemic pregnant women will develop an aquatic physical exercise in a thermal pool, 45 minutes per one time, from rehabilitation center of the IMIP. Before to practice the aquatic exercise women will have their physical capacity assessed by the Six minutes walk test and fetal conditions will be assessed by ultrasound. They will also be submitted to a dermatological examination by specialist. Primary endpoint will be glucose levels (glycemic test), secondary endpoints will be the following maternal and fetal: blood pressure, heart rate, respiratory rate, oxygen saturation level, fetal cardio beat and fetal movement.The variables will be measured before and after the water exercise session. Maternal and fetal characteristics of the study sample will be presented by group, intervention and control in terms of mean and standard deviation. For group comparisons of glucose levels and maternal and fetal variables, continuous and nominal data will be analyzed by t test for unpaired data and χ2 tests, respectively. Data will be analyzed using the intention-to-treat principle. Statistical analysis will be performed with the STATA version 12.0 and the level of significance will set to <0.05. Even in cases where there is the appearance of some criterion for discontinuation during the intervention (Aquatic physical exercise), the patient will be considered part of the group which was initially included in the randomization (intent to treat) and is not excluded from the study. The physical proprieties of water provide aquatic exercises as ideal for pregnant women. An aquatic physical exercise program developed with pregnant women in a thermal pool and under a physiotherapist supervision must ensure compliance. It is expected that this study provide evidences to the real role of aquatic physical exercise on glycemic control of GDM.

ELIGIBILITY:
Inclusion Criteria:

* GDM Group: GDM diagnosis will be based on International Association of the Diabetes in Pregnancy Study Group (IADPSG) and WHO, Hyperglycemia and Adverse Pregnancy Outcomes (HAPO) study (2 h 75 g oral glucose tolerance test (OGTT): a fasting glucose ≥ 92 mg/dl or a one hour result of ≥ 80 mg/dl, or a two hour result of ≥ 153 mg/dl;
* Control Group: Normal glucose tolerance (IADPSG /WHO)
* Aging 18 to 35 years;
* Physically inactive (< 150' per week based on International Physical Activity Questionnaire.

Exclusion Criteria:

* Kidney disease or collagenosis;
* Previous history of gestational diabetes;
* Diabetes type 1 or type 2;
* Hypertensive disorders related to pregnancy;
* Hemodynamic instability;
* Obstetric labor;
* Vaginal bleeding;
* Cognitive disorder, auditory, visual or motor severely limiting, attested by a medical specialist;
* Skin disorders who have a contraindication to the use of a swimming pool;
* Urinary tract infection;
* Be inserted in the program of regular exercise;

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-03; Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change from Glycemic level | Before and up to 5 minutes after the intervention
  Blood glucose test: maternal glucose levels

SECONDARY OUTCOMES:
Change from Systolic and diastolic blood pressure | Before and up to 5 minutes after the intervention
  Measured in mmHg every medical consultation
Change from Heart rate (pulse) | Before and up to 5 minutes after the intervention
  number of beats in 60 seconds
Change from Respiratory rate | Before and up to 5 minutes after the intervention
  number of movements indicative of inspiration and expiration per 60 seconds
Change from Oxygen saturation | Before and up to 5 minutes after the intervention
  Quantity oxygen is being transported in the blood at the time of measurement
Change from Fetal heart rate | Before and up to 5 minutes after the intervention
  Heartbeat frequency of the fetus per minute

CONTACTS AND LOCATIONS:
Overall Officials: João Guilherme Bezerra Alves/, Doctor, Study Director — Institute of Integrative Medicine Professor Fernando Figueira; Alex Sandro Rolland de Souza, Doctor, Study Chair — Institute of Integrative Medicine Professor Fernando Figueira
Locations (1):
- José Roberto da Silva Junior, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No